CLINICAL TRIAL: NCT03604107
Title: Evaluation of the Efficacy of Preimplantation Genetic Screening (PGS) in Predicting Embryonic Ploidy and Subsequent Pregnancy Outcomes in in Vitro Fertilization (IVF) Cycles
Brief Title: Predictive Value of Embryonic Testing
Acronym: PROV-ET
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2018-01
Record Dates: First submitted 2018-06-14; First posted 2018-07-27 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, buccal swab, rectal/vaginal swab, endometrial biopsy and aspirate, discarded specimens leftover after an IVF procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Preimplantation Genetic Testing-Aneuploidy — trophectoderm biopsy samples will be analyzed for karyotype after clinical outcome is determined

SUMMARY:
The primary objective of this study is to determine the predictive value of preimplantation genetic screening (PGS) as a marker of embryonic competence. Secondary objectives are to define the related or independent predictive values of other proposed markers of embryonic and maternal reproductive competence in assisted reproductive technology (ART) cycles.

DETAILED DESCRIPTION:
Patients participating in the study will undergo a routine in vitro fertilization cycle. Trophectoderm biopsy will be performed on all blastocysts however biopsy samples will not be analyzed till the clinical outcome has been determined. The single, morphologically best embryo available will be selected for transfer. All clinical and laboratory care is identical to that of which subjects would receive if they were not participating in the study. This includes all pretreatment screening, in-cycle treatment, embryology procedures, single embryo transfer, pregnancy testing, and pregnancy follow-up (if pregnancy occurs).

ELIGIBILITY:
Inclusion Criteria:

1. Couples electing embryonic aneuploidy screening (PGS)
2. Couples electing single embryo transfer

Exclusion Criteria:

1. Any prior failed IVF cycle
2. Diagnosis of endometrial insufficiency: prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), persistent endometrial fluid
3. Diagnosis of chronic endometritis
4. Maximum day 3 FSH level of 12 or higher
5. Anti-mullerian hormone level less than 0.5 g/mL, tested within previous year
6. Total basal antral follicle count less than 8 follicles
7. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
8. BMI <18.5 or > 35
9. Personal history of recurrent pregnancy loss (two or more pregnancy losses)
10. Use of oocyte donation
11. Use of gestational carrier
12. Medical condition predisposing patient to high risk pregnancy
13. Use of surgical procedures to obtain sperm
14. Presence of hydrosalpinges that communicate with endometrial cavity
15. Any contraindications to undergoing in vitro fertilization or gonadotropin stimulation
16. Single gene disorder or chromosomal rearrangement requiring a more detailed embryonic genetic analysis

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Infertile couples attempting conception through in vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Predictive Value of Aneuploidy Screening | approximately 1 month post clinical outcome
  Determine confidence intervals that a euploid embryo will implant, an aneuploid embryo will not implant, and the likelihood of mosaic and segmental aneuploid embryos implanting and describe their outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott Jr., MD, HCLD, Principal Investigator — IVI RMA
Locations (4):
- United States (4):
  - Reproductive Medicine Associates of Florida, Lake Mary, Florida
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reproductive Medicine Associates of Pennsylvania, Allentown, Pennsylvania
  - Reproductive Medicine Associates of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiegs AW, Tao X, Zhan Y, Whitehead C, Kim J, Hanson B, Osman E, Kim TJ, Patounakis G, Gutmann J, Castelbaum A, Seli E, Jalas C, Scott RT Jr. A multicenter, prospective, blinded, nonselection study evaluating the predictive value of an aneuploid diagnosis using a targeted next-generation sequencing-based preimplantation genetic testing for aneuploidy assay and impact of biopsy. Fertil Steril. 2021 Mar;115(3):627-637. doi: 10.1016/j.fertnstert.2020.07.052. Epub 2020 Aug 28. PMID 32863013